CLINICAL TRIAL: NCT04826705
Title: A Prospective, Multicenter, Observational Study of Short and Long-term Outcome in Endovascular Treatment of Femoropopliteal Arterial Occlusive Lesion With Drug-Coated Balloon (PROMISING Study)
Brief Title: A Study of Endovascular Treatment of Femoropopliteal Arterial Occlusive Lesion With Drug-Coated Balloon
Acronym: PROMISING
Status: Active, not recruiting | Type: Observational
Sponsor: Liyuan Hospital of Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: RenJi Hospital (Other); Zhejiang University (Other); Xuanwu Hospital, Beijing (Other); First People's Hospital of Hangzhou (Other); Second Affiliated Hospital of Suzhou University (Other); Qingdao University (Other); Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Zibo Feng, Director of Vascular Surgery, Liyuan Hospital, Liyuan Hospital of Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: the PROMISING Study
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2023-12

CONDITIONS: Drug-coated Balloon; Femoropopliteal Artery Occlusion; Angioplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Drug-coated Balloon — To observe the effectiveness and safety of the drug-coated balloon in the treatment of lower extremity arteriosclerosis obliterans of the femoral popliteal artery segment.

SUMMARY:
There have been a number of randomized controlled studies (RCT) showing the efficacy of the endovascular treatment with drug-coated balloons (DCB) in the femoropopliteal artery lesions. However, these studies have been carefully designed, and most of them have excluded long-length lesions and severely calcified lesions. In addition to being used alone in the real word, drug-coated balloons (DCB) are also used in combination with stents or debulking devices, but in these randomized controlled studies (RCT) they are only compared with standard percutaneous transluminal angioplasty (PTA). Therefore, the investigators initiated this study, which is a prospective, multicenter, observational real-world study of short and long-term outcome in endovascular treatment of femoropopliteal arterial occlusive lesions with DCB.

DETAILED DESCRIPTION:
Traditional endovascular approaches to the treatment of atherosclerotic disease in the femoropopliteal arteries include percutaneous transluminal angioplasty (PTA) with an uncoated balloon and implantation of a bare metal stent. Recently, drug-eluting stents (DES) and drug-coated balloons (DCB) that transfer paclitaxel to the vessel wall during revascularization have been added to the suite of tools available to interventionists, helping to prevent restenosis after treatment.

There have been a number of randomized controlled studies (RCT) showing the efficacy of the endovascular treatment with drug-coated balloons (DCB) in the femoropopliteal artery lesions. However, these studies have been carefully designed, and most of them have excluded long-length lesions and severely calcified lesions. In addition to being used alone in the real word, drug-coated balloons (DCB) are also used in combination with stents or debulking devices, but in these randomized controlled studies (RCT) they are only compared with standard percutaneous transluminal angioplasty (PTA).

Therefore, the investigators initiated this study, which is a prospective, multicenter, observational real-world study of short and long-term outcome in endovascular treatment of femoropopliteal arterial occlusive lesions with DCB. It is estimated that 1200 patients with chronic femoral popliteal artery occlusion were enrolled in the group at 8 centers in China in two years. The follow-up would be conducted at 1, 3, 6, 12, 18, 24, 36 and 48 months after the operation to assess the efficacy and safety of the endovascular treatment with drug-coated balloons (DCB) in the femoropopliteal artery lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Rutherford grade 2-5.
2. Femoral popliteal artery stenosis or occlusion, a clear outflow tract no less than 10cm long at the distal end of the knee should be continuous with a clear outflow tract under the ankle.
3. Patients who understand the purpose of this study, volunteer to participate in the experiment, sign informed consent and are willing to follow up.
4. The guide wire needs to pass through the lesion.
5. Life expectancy> 24 months.
6. Patients with thrombosis of the lower extremities, patients who received drug-coated balloon (DCB) intervention after thrombus removal through mechanical thrombus removal, percutaneous catheter thrombolysis, and thrombus removal.
7. Patients who have received DCB intervention for both lower limbs can be enrolled in the group according to the intracavitary treatment time.
8. There is at least one continuous infrapopliteal outflow artery or obtained through intravascular reconstruction.
9. For combined aortic iliac artery disease, the blood flow can be recanalized after intravascular reconstruction without residual stenosis exceeding 50%.

Exclusion Criteria:

1. Patients with stroke, cerebral hemorrhage, gastrointestinal hemorrhage or myocardial infarction within 3 months before enrollment.
2. Patients who are known to be allergic to heparin, aspirin, other antiplatelet drugs, contrast agents, etc.
3. Patients who have participated in clinical trials of drugs or other medical devices that interfere with this clinical trial within the past 3 months.
4. Pregnant and lactating women.
5. Patients who are unable or unwilling to participate in this trial.
6. Patients with Berg's disease.
7. Patients who have undergone arterial bypass on the treatment side.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with femoralpopliteal artery occlusion.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from clinically-driven target lesion revascularization(CD-TLR) rate at post-interventional | 48 months
  Clinically-driven target lesion revascularization (CD-TLR) is defined as any re-intervention within the target lesion due to symptoms or drop of ankle brachial index (ABI) of ≥20% or >0.15 when compared to post-procedure baseline.
Major adverse events | 48 months
  Operation-related acute thrombosis, arterial embolism, major amputation and all-cause mortality.

SECONDARY OUTCOMES:
Changes of the patency rate of target lesions at post-interventional | 1 month, 3 months, 6 months, 12 months, 24 months, 36 months, 48 months
  The patency rate of target(Femoropopliteal) lesions would be determined by vascular ultrasound,Restenosis would be diagnosed if the peak systolic velocity ratio(PSVR)≥2. 5.
Technical success rate | 1 week
  Successfully revascularize the target vessel. The residual stenosis is <30% and there is no acute thrombosis occurred in the target vessel within 1 week post-operation.
Vascular quality of life questionnaire(VascuQol) | 1 month, 3 months, 6 months, 12 months, 24 months, 36 months, 48 months
  The VascuQol was designed as a questionnaire containing five domains: pain (4 items), symptoms (4 items), activities (8 items), social (2 items), and emotional (7 items) to evaluate Health related quality of life (HRQL). Every item has seven response options, with scores ranging from 1 to 7. A total score is the sum of all 25 item scores divided by 25.And both the total score as well as the domain scores range from 1 (worst HRQL) to 7 (best HRQL).The lower the value, the poorer the quality of life.
The patient's ulcer healing | 1 month, 3 months, 6 months, 12 months, 24 months, 36 months, 48 months
  Ulcer healing in patients with Rutherford grade 5
Freedom from clinically-driven target lesion revascularization(CD-TLR) rate at post-interventional | 1 month, 3 months, 6 months, 12 months, 24 months, 36 months
  Clinically-driven target lesion revascularization (CD-TLR) is defined as any re-intervention within the target lesion due to symptoms or drop of ankle brachial index (ABI) of ≥20% or >0.15 when compared to post-procedure baseline.
Major adverse events | 1 month, 3 months, 6 months, 12 months, 24 months, 36 months
  Operation-related acute thrombosis, arterial embolism, major amputation and all-cause mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Zibo Feng, Principal Investigator — Liyuan Hospital of Tongji Medical College, Huazhong University of Science and Technology
Locations (9):
- China (9):
  - Zibo Feng, Wuhan, Hubei
  - Xuanwu Hospital Capital Medical University, Beijing
  - Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu
  - Hangzhou First People's hospital of Medical College of Zhejiang University, Hangzhou
  - the First Affiliated hospital of Medicine College of Zhejiang University, Hangzhou
  - Qingdao Haici hospital affiliated to Qingdao University, Qingdao
  - Renji Hospital of Shanghai Jiaotong University, Shanghai
  - Zhongshan Hospital of Fudan University, Shanghai
  - the second Affiliated Hospital of Medical College of Suzhou University, Suzhou

IPD SHARING:
Plan to Share IPD: Undecided
Share data with multi-center participants in this study.